CLINICAL TRIAL: NCT05271084
Title: Pentoxifylline as an Adjunct to Citalopram in Adult Patients With Major Depressive Disorder: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Pentoxifylline as an Adjunct to Citalopram in Adult Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Talar A. Merza Mohammad, Associate Professor of Department of Pharmacology and Toxicology, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMU PE-EC 16112021/382
Record Dates: First submitted 2022-02-23; First posted 2022-03-08 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Citalopram; Tablets; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citalopram + Pentoxifylline group (Experimental): Citalopram (tablet): 20 mg once a day for 12 weeks + Pentoxifylline (tablet): 400 mg twice a day for 12 weeks
  Interventions: Drug: Citalopram (tablet) 20 mg + Pentoxifylline (tablet) 400Mg
- Control group (Placebo Comparator): Citalopram (tablet): 20 mg once a day for 12 weeks + placebo (tablet) twice a day for 12 weeks
  Interventions: Drug: Citalopram (tablet) 20 mg + Placebo (tablet)

INTERVENTIONS:
Drug: Citalopram (tablet) 20 mg + Pentoxifylline (tablet) 400Mg — Selective serotonin reuptake inhibitor (SSRI) + phosphodiesterase inhibitor with anti-inflammatory properties
  Arms: Citalopram + Pentoxifylline group
Drug: Citalopram (tablet) 20 mg + Placebo (tablet) — Selective serotonin reuptake inhibitor (SSRI) + placebo
  Arms: Control group

SUMMARY:
The aim of this study is to test if combining the antidepressant Citalopram with Pentoxifylline (PTX), a medicine with anti-inflammatory and phosphodiesterase inhibitory properties, enhanced antidepressant efficacy in adult patients with major depressive disorder (MDD) when compared to Citalopram alone.

DETAILED DESCRIPTION:
According to mounting evidence, inflammation and phosphodiesterase (PDE) pathways may play a role in the pathogenesis of psychiatric diseases such as MDD. PTX is a phosphodiesterase inhibitor and has anti-inflammatory and antioxidant effects. Therefore, it has been hypothesized that MDD patients taking combined administration of the Citalopram, a Selective Serotonin Reuptake Inhibitor (SSRI), and PTX would show a higher improvement in depression symptoms. The relationship between the Hamilton Depression Rating Scale-17 items (Ham-D-17) score and various biological markers and their potential role in the therapeutic outcome of MDD will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, voluntary informed consent prior to study enrollment.
* Male or female between the ages of 21 to 65.
* Patient must be diagnosed with a moderate to a severe depressive episode, as determined by the MADRS score >21.
* Prior to taking part in the trial, all patients were requested to abstain from all psychotropic and anti-inflammatory medications for at least four weeks.

Exclusion Criteria:

* Current psychotic symptoms or perceptual problems of any kind, at the discretion of the investigator
* The presence of a contraindication to PTX, such as a drug allergy or xanthine derivative allergy
* The presence of cardiovascular diseases, including high blood pressure, a recent myocardial infarction, cardiac arrhythmia, coronary artery disease, or a coagulation disorder
* Renal impairment, defined as creatinine clearance less than 80ml/min
* Patients who have previously received electroconvulsive therapy (ECT)
* Patients who have inflammatory disorders
* Patients with a concurrent active medical condition
* Patients with a history of seizures
* Patients who are pregnant or nursing females.
* Patients with bipolar I or bipolar II disorder
* Patients with personality disorders
* Patients with eating disorders
* Patients with substance dependence or abuse

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale 17 (HDRS-17) Scores (Time Frame: Baseline, week 2,4,6,8,10, and12) | 12 weeks
  The HDRS is a 17-item scale that asks participants to rate the severity of their depression symptoms. Scoring is based on the 17-item scale. The total score ranges from 0 to 52, with higher numbers demonstrating more severe symptoms. Normal scores range from 0 to 7, mild depression ranges from 8 to 16, moderate depression ranges from 17 to 23, and scores of 24 and greater indicate severe depression. Remission is defined as HDRS total score ≤ 7 (primary outcome).

SECONDARY OUTCOMES:
Effect on the serum level of tumor necrosis factor-alpha (TNF-α) | 12 weeks
  Peripheral blood samples will be obtained and serum levels of TNF-α ( pg/mL) will be measured at baseline and after treatment (week 12)
Effect on the serum level of circulating C-reactive protein (CRP) | 12 weeks
  Peripheral blood samples will be obtained and serum levels of CRP (mg/dL) will be measured at baseline and after treatment (week 12)
Effect on the serum level of interleukin 6 (IL-6) | 12 weeks
  Peripheral blood samples will be obtained and serum levels of IL-6 (pg/mL) will be measured at baseline and after treatment (week 12)
Effect on the serum level of interleukin-1-β (IL-1-β) | 12 weeks
  Peripheral blood samples will be obtained and serum levels of IL-1-β (pg/mL) will be measured at baseline and after treatment (week 12)
Effect on the serum level of interleukin-10 (IL-10) | 12 weeks
  Peripheral blood samples will be obtained and serum levels of IL-10 (pg/mL) will be measured at baseline and after treatment (week 12)
Effect on the serum level of brain derived neurotrophic factor (BDNF) | 12 weeks
  Peripheral blood samples will be obtained and serum levels of BDNF (ng/mL) will be measured at baseline and after treatment (week 12)
Effect on the serum level of serotonin | 12 weeks
  Peripheral blood samples will be obtained and serum levels of serotonin (ng/mL) will be measured at baseline and after treatment (week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Talar A Merzamohammad, Pharm. D, Principal Investigator — Hawler Medical University, College of Pharmacy, Department of Pharmacology and Toxicology
Locations (1):
- Hawler Psychiatric Hospital and Private Clinic, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No